CLINICAL TRIAL: NCT01268293
Title: A Phase 1 Study of E7080 in Subjects With Solid Tumor
Brief Title: A Study of E7080 in Subjects With Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-J081-105
Record Dates: First submitted 2010-12-28; First posted 2010-12-30 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2016-08

CONDITIONS: Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasms | interventions — lenvatinib

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E7080

INTERVENTIONS:
Drug: E7080 — This arm will be a dose-escalation evaluation of 9-18 subjects to investigate the tolerability and safety of E7080 up to 24 mg when administered orally on a once daily continuous dose schedule in cycles (4 weeks as 1 cycle). Administration of the study drug can continue until subjects meet discontinuation criteria such as disease progression, intolerable toxicity, and withdrawal of study consent.

SUMMARY:
The purpose of this study is to investigate the tolerability and safety of E7080 up to 24 mg when administered orally on a once daily continuous dose schedule in cycles (4 weeks as 1 cycle) in subjects with solid tumors

ELIGIBILITY:
Inclusion Criteria

* Subjects with histologically and/or cytologically diagnosis of solid tumor
* Subjects with solid tumor which is resistant to standard anti-tumor therapies, or which no appropriate treatment is available
* Subjects whose toxicity of previous treatment has recovered to Grade 1 or lower toxicity (except for alopecia)
* Subjects who completed previous anti-tumor therapy before at least 4 weeks
* Subjects who are 20 years or older
* Subjects with 0 to 1 of Performance Status
* Subjects agree to be hospitalized for DLT observation
* Subjects with adequate organ functions
* Males and females of childbearing potential must agree to use appropriate contraception from the agreement to 30 days after study drug administration.
* Agree to participate in this study in writing based on voluntary will

Exclusion Criteria

* Subjects with brain metastasis accompanying clinical symptoms or requiring treatment
* Subjects with the severe complication or disease history
* Subjects unable to take oral medication.
* Subjects being treated with drugs that strongly inhibit or induce CYP3A4 and that may be possibly used during this study.
* Scheduled for surgery during the projected course of the study.
* Positive for human immunodeficiency virus (HIV antibody) test or positive for hepatitis B surface (HBs antigen) or hepatitis C (HCV antibody) by serum test.
* Subjects who in the view of the investigator are not able to comply with this protocol because of psychiatric or physical diseases including alcoholism or drug addict
* Pregnant or nursing subjects
* Subjects who are participating in another clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuya Sasaki, Study Director — Oncology Clinical Development Section. JAC PCU. Eisai Co., Ltd.
Locations (1):
- Chuo-ku, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- E7080: E7080 was administered orally once day (QD) in the morning. The initial dose of E7080 was 20 mg QD and increased to 24 mg QD if 20 mg was confirmed to be tolerable.
Period: Overall Study
Arm/Group | E7080
Started | 9
Completed Cycle 1 | 9
Completed | 0
Not Completed | 9
Not completed — Disease progression | 7
Not completed — Adverse Event | 1
Not completed — Subject choice | 1

BASELINE CHARACTERISTICS:
Arm/Group | E7080
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.6 (11.5)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 2
  Female | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Time Frame: Up to 4 weeks
Population: Subjects with less than 75% compliance in Cycle 1 for reasons other than the toxicity of the study drug and who discontinued prior to confirmation of tolerability in Cycle 1 were excluded from the analysis of DLT. All 9 participants completed Cycle 1 (DLT monitoring period) and were included in the analysis of DLT.
Measure: Number; unit: Participants
Arm/Group | E7080
Number analyzed (Participants) | 9
Participants | 0

2. Primary Outcome: Number of Participants With Adverse Events
Description: Treatment emergent adverse events (AEs) and serious adverse events (SAEs) were evaluated by determining the AE grade according to Common Terminology Criteria for Adverse Events [CTCAE] version 4.0, laboratory tests, vital signs (blood pressure [mm Hg], heart rate [beats per minute], body temperature [degree C], and body weight [kg]), 12-lead electrocardiograms (ECGs; heart rate [bpm], QT [msec] and QTc [msec]) and Eastern Cooperative Oncology Group performance status (ECOG-PS).
Time Frame: Until participants met discontinuation criteria such as disease progression, intolerable toxicity, and withdrawal of study consent or up to 19 cycles (1 cycle = 28 days).
Population: The Safety Analysis Set consisted of subjects who had received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Measure: Number; unit: Participants
Arm/Group | E7080
Number analyzed (Participants) | 9
Participants | 9

ADVERSE EVENTS:
Time Frame: Until participants met discontinuation criteria such as disease progression, intolerable toxicity, and withdrawal of study consent or up to 19 cycles (1 cycle = 28 days).
Arm/Group | E7080
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E7080 (N=9)
Diarrhoea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E7080 (N=9)
Anaemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 7
Lymphopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Hyperthyroidism (Endocrine disorders) | 3
Hypothyroidism (Endocrine disorders) | 3
Eye pruritus (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Malaise (General disorders) | 6
Oedema peripheral (General disorders) | 4
Pyrexia (General disorders) | 2
Cystitis (Infections and infestations) | 2
Infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Paronychia (Infections and infestations) | 2
Wound complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 6
Blood alkaline phosphatase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 6
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 4
Blood thyroid stimulating hormone increased (Investigations) | 8
Blood urine present (Investigations) | 1
Electrocardiogram T wave inversion (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 2
Occult blood (Investigations) | 1
Urine ketone body present (Investigations) | 1
Weight decreased (Investigations) | 2
Weight increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Hyperchloraemia (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4
Hypoproteinaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 7
Insomnia (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 4
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other